CLINICAL TRIAL: NCT00060099
Title: Phase II Randomized, Double-Blinded Trial Of SGN-00101 (HSP-E7) For Treatment Of CIN II/III
Brief Title: SGN-00101 in Treating Patients With Cervical Intraepithelial Neoplasia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dana-Farber/Brigham and Women's Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: CDR0000299462; BWH-000-P-CONS01; NCI-3074
Record Dates: First submitted 2003-05-06; First posted 2003-05-07 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2005-03

CONDITIONS: Precancerous Condition
Keywords: cervical intraepithelial neoplasia grade 2; cervical intraepithelial neoplasia grade 3; human papilloma virus infection
MeSH Terms: conditions — Precancerous Conditions; Uterine Cervical Dysplasia; Papillomavirus Infections

INTERVENTIONS:
Biological: HspE7

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development of or treat early cancer. SGN-00101 may be effective in preventing the development of cervical cancer in patients with cervical intraepithelial neoplasia.

PURPOSE: This randomized phase II trial is studying how well SGN-00101 works in preventing cervical cancer in patients with cervical intraepithelial neoplasia and human papillomavirus.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of SGN-00101 vs placebo in patients with grade II or III cervical intraepithelial neoplasia.
* Correlate clinical response, as defined by histologic demonstration of lesion regression, with potential surrogate markers of vaccine efficacy (e.g., spectroscopic changes in the epithelium, development of human papilloma virus (HPV)-specific mucosal and systemic T-cell responses, and levels of HPV-specific antibody in cervical secretions), in patients treated with this drug.

OUTLINE: This is a randomized, double-blind study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive SGN-00101 subcutaneously (SC) once a month for 3 consecutive months in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive placebo SC as in arm I. Patients are followed monthly for 3 months after the last injection and then undergo large loop excision of the transformation zone under colposcopy at the fourth month. Patients with disease progression undergo immediate large loop excision.

PROJECTED ACCRUAL: A maximum of 80 patients (40 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed grade II or III cervical intraepithelial neoplasia

  * Confirmed by colposcopy-directed punch biopsy
* Accessible, definable, and entirely visible cervical lesions persisting after biopsy

  * Satisfactory colposcopic exam within 3-6 weeks after diagnostic biopsy
* Positive for human papilloma virus 16
* CD4+ counts normal

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0

Life expectancy

* Not specified

Hematopoietic

* No coagulation disorder that requires medical intervention

Hepatic

* Hepatitis B core antigen negative
* Hepatitis C antibody negative

Renal

* Not specified

Cardiovascular

* No cardiovascular disorder that requires medical intervention

Pulmonary

* No respiratory disorder that requires medical intervention

Immunologic

* HIV negative
* Not immunologically compromised
* No prior severe allergic reactions (anaphylactic response) to drugs or any other allergen
* No immunological disorders including any of the following:

  * Lupus
  * Diabetes
  * Multiple sclerosis
  * Myasthenia gravis
* No active systemic infections that require medical intervention

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Willing to undergo a loop electrosurgical excision procedure
* No medical or psychiatric illness that would preclude study treatment, ability to give informed consent, or study compliance
* No other prior malignancy except nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent immunotherapy
* No other concurrent gene therapy
* No concurrent biologic therapy

Chemotherapy

* No concurrent chemotherapy

Endocrine therapy

* More than 30 days since prior systemic steroid therapy

Radiotherapy

* No concurrent radiotherapy

Surgery

* Not specified

Other

* More than 30 days since prior investigational drugs
* No other concurrent investigational drugs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-05

CONTACTS AND LOCATIONS:
Overall Officials: Kristin A. Keefe, MD, Study Chair — Dana-Farber/Brigham and Women's Cancer Center
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States